CLINICAL TRIAL: NCT02991950
Title: Weight Adjusted Low Molecular Weight Heparin in Recurrent Implantation Failure: a Randomized Open Labeled Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty with patient enrollment
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 876
Record Dates: First submitted 2016-11-29; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Infertility; Low Molecular Weight Heparin
MeSH Terms: conditions — Infertility | interventions — parnaparin; Fluxum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parnaparin sodium (Experimental): Women in LMWH arm are administered with routine ovulation induction protocol and prophylactic dose of parnaparin sodium (LMWH), starting the day before the beginning of stimulation phase of the cycle until the result of the procedure is confirmed in terms of pregnancy yes or no and in case of pregnancy until the delivery or the end of pregnancy. Women in the LMWH arm will be tested for blood cell count twice in the first 10 days of therapy.
  Parnaparin will be administered at the dose of 100 IU/kg/day from the day before the beginning of stimulation phase of the cycle until the result of the procedure is confirmed in terms of pregnancy yes or no and in case of pregnancy until delivery or the end of the pregnancy.
  Used dosages Parnaparin 0.4 4250 UI Parnaparin 0.6 6400 UI
  Interventions: Drug: Parnaparin Sodium
- no treatment (No Intervention): Women in the control arm are administered with routine ovulation induction protocol, without the addition of parnaparin sodium.

INTERVENTIONS:
Drug: Parnaparin Sodium — Parnaparin sodium ( Fluxum 4250 anti-Xa IU /0.4 mL or Fluxum 6400 anti-Xa IU /0.6mL; Alfa Wassermann S.p.A.) was administered at a dose of 100 IU/kg/day from the day before the beginning of the stimulation phase of the cycle until the result of the procedure was confirmed by pregnancy and, in the case of evolutive pregnancy, until delivery or the end of pregnancy
  Other Names: Fluxum
  Arms: parnaparin sodium

SUMMARY:
Prospective randomized study of patients with infertility candidates to Assisted ReproductiveTechniques (ART), screened for all inclusion and exclusion criteria, submitted to ART cycle with or without low molecular weight heparin (LMWH) administration. Aims of the study are to evaluate, primarily, pregnancy rate/embryo transfer, secondarily take home babies/embryo transfer, implantation rate, and the role of thrombophilic factors

DETAILED DESCRIPTION:
This is an interventional, stratified, randomized, open blind study. It will conducted on outpatients selected on the basis of inclusion and exclusion criteria.

Patients will be randomised according to a computer generated list of randomization to receive or not LMWH at prophylactic daily dosage (100 IU/kg).

For a correct selection and analysis some parameters have to be checked before randomization (see randomization check list at the end). The women in LMWH arm will treated starting the day before the beginning of stimulation phase of the cycle of ART until the result of the procedure is confirmed in terms of pregnancy yes or no, and if the pregnancy will be confirmed until the delivery or the end of pregnancy. Women in the control arm are administered routine hormonal support without LMWH.

Data will be collected on smoking habits, BMI, the number of retrieved oocytes, transferred embryos and implantation rate, ART outcome and parameters used for randomization on the basis of inclusion and exclusion criteria.

During the study blood will be collected for analysis at the randomization, the moment in wich patient will be assigned to one of the two arms, at the transfer and at the day of check for betaHCG and in in case of pregnancy all women will be checked at 12, 24, 36 week for testing of functional parameters of coagulation (protein C, protein S, AT, ddimer, fibrinogen, PT, aPTT, FVII, FVIII, FIX, and vonWillebrand factor antigen), blood cells count and of lipids (cholesterol and triglycerides).

The samples, identified with a sequential identification number, will be collected, processed and storage at -20/-80°C in the promoter center and will be destroyed after the analyses.

Study treatment Women in LMWH arm are administered with prophylactic weight adjusted dose of LMWH, starting the day before the beginning of stimulation phase of the cycle until the result of the procedure is confirmed in terms of pregnancy yes or no and in case of pregnancy until the delivery or the end of pregnancy. Women in the LMWH arm will be tested for blood cell count twice in the first 10 days of therapy.

Initial dose and schedule Parnaparin will be administered at the dose of 100 IU/kg/day from the day before the beginning of stimulation phase of the cycle until the result of the procedure is confirmed in terms of pregnancy yes or no and in case of pregnancy until delivery or the end of the pregnancy.

None of patients can receive concomitant acetylsalicylic acid (ASA) or steroids therapy Treatment duration

Women in LMWH arm are administered with prophylactic weight adjusted dose of parnaparin, starting the day before the beginning of stimulation phase of the cycle until the result of the procedure is confirmed in terms of pregnancy yes or no and in case of pregnancy until the delivery or the end of the pregnancy.

Whatever the disease status, the treatment will always be discontinued in case of patient refusal excessive toxicity precluding further therapy, according to the responsible physicianother complications, according to the responsible physician

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years and ≤40 years, candidated to a fresh IVF/ICSI cycle with routine ovulation induction protocol

Exclusion Criteria:

v-vCouples candidated to a frozen IVF/ICSI cycle with routine ovulation induction protocol

* Testicular or frozen sperm (TESE procedure not allowed)
* Presence of hormonal disorders not compensated with specific therapy or history of immunological disease (autoimmune thyroiditis, connectivitis, RA, SLE, etc )
* Presence of antiphospholipides autoantibodies or other severe thrombophilia (AT, PS, PC deficiency or homozygous FV Leiden or FIIG20210A, or double eterozygous FV Leiden and FIIG20210A)
* Presence of abnormal platelets count and congenital or acquired coagulopathy ASA or steroid therapy administration

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2011-07; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pregnancy rate/embryo transfer | 12-14 days
  the investigators measured the pregnancy rate/embryo transfer using betaHcg dosage 12 days after embryo transfer

SECONDARY OUTCOMES:
take home babies/embryo transfer | 38-40 weeks after embryo transfer
  Live birth was defined as delivery of one or more live infants after 23 gestational weeks.
implantation rate | 3 weeks
  ultrasound was performed to evaluate implantation rate calculated as as number of gestational sacs divided by number of transferred embryos multiplied by 100
role of thrombophilia in interfering with pregnancy rate/take home baby/implantation rate | 12-14 days and 38-40 weeks and 3 weeks
  All enrolled patients were previously screened for the presence or not of thrombophilic defects: protein C or protein S or AT deficiency, FV G1691A and FIIG20210A mutations, C677T MTHFR polymorphism,hyperhomocysteinemia, antiphospholipid antibodies. The investigators excluded from the enrollment patients with severe thrombophilia: protein C, protein S, AT deficiency or homozygous FV Leiden and FIIG20210A mutations or double heterozygosity for FV Leiden and FIIG20120 mutations because in this patients the international guide lines suggest and recommend the use of antithrombotic prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: corrado lodigiani, MD,PHD, Principal Investigator — Thrombosis Center

IPD SHARING:
Plan to Share IPD: No